CLINICAL TRIAL: NCT03008538
Title: Dental Implant Placement in Extraction Socket of Mandibular Anterior and Premolar Areas Treated With Mineralized Plasmatic Matrix Versus Autogenous Bone Graft
Brief Title: Socket Preservation Using Autogenous Bone Graft Versus MPM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khaled Jamal Taha Hussien, Dentist Msc, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CairoSPR-Aut
Record Dates: First submitted 2016-12-26; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Bone Graft; Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mineralized Plasmatic Matrix (Experimental): MPM(Mineralized plasmatic matrix) insertion in extraction sockets for socket preservation for later implant placement and histomorphometric analysis.
  Interventions: Other: MPM(Mineralized plasmatic matrix).
- Autogenous Bone Graft (Gold Standards). (Active Comparator): Socket preservation using Autogenous bone graft for later implant placement and histomorphometric analysis.
  Interventions: Other: Autogenous Bone Graft

INTERVENTIONS:
Other: MPM(Mineralized plasmatic matrix). — Preparation of sticky bone graft by addition of growth factors obtained from patient's vebous blood.
  Other Names: Sticky bone graft.
  Arms: Mineralized Plasmatic Matrix
Other: Autogenous Bone Graft — Socket preservation using autogenous bone graft for preservation of bone width and height for future implant insertion.
  Other Names: Gold Standards
  Arms: Autogenous Bone Graft (Gold Standards).

SUMMARY:
Studying the comparative effectiveness of socket preservation using autogenous bone graft versus MPM for implant insertion.

DETAILED DESCRIPTION:
To assess bone quality, stability of implants placed in fresh extraction sockets of mandibular anterior and premorals augmented by MPM (Mineralized Plasmatic Matrix) versus autogenous bone graft (gold standard), at different follow-up periods (0, 3, 6, 9 months).

ELIGIBILITY:
Inclusion Criteria:

1. Medically free patients.
2. Patients with mandibular anterior and premolar hopeless teeth indicated for extraction.
3. Evaluated bone height on X.Ray to be (0-4 mm buccal bone dehiscence).
4. Age between 18 and 40 years.
5. Both sexes.
6. Patients physically able to tolerate surgical and restorative procedures. Good oral hygiene.
7. Highly motivated patients.

Exclusion criteria:

1. Smokers.
2. Pregnant or lactating females.
3. Presence of any pathosis in the pre-implant site.
4. Presence of Para functional habits.
5. History of oral radiotherapy.
6. History of prolonged steroids use
7. Psychological disorders.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction regarding function, to be measured using patient questionnaire. | 3 Months.

SECONDARY OUTCOMES:
Comparative histomorphometric analysis, to be measured using a digital software called (leica QWin 500) and unit of measurements are to be (Pixels). | 3 Months.

IPD SHARING:
Plan to Share IPD: Undecided